CLINICAL TRIAL: NCT01933464
Title: An Analysis of the Effect of Topical Cromolyn Sodium on Rosacea-associated Erythema
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Anna Di Nardo, MD, PhD, MD, PhD (Associate Professor of Medicine), University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 130199
Record Dates: First submitted 2013-08-21; First posted 2013-09-02 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-07

CONDITIONS: Papulopustular Rosacea
Keywords: Rosacea; Cromolyn sodium
MeSH Terms: conditions — Rosacea | interventions — Cromolyn Sodium; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cromolyn (Experimental): Subjects in this arm will be asked to apply their assigned medication twice daily to their entire face. The medication they will be receiving is cromolyn sodium ophthalmic solution, 4%.
  Interventions: Drug: Cromolyn Sodium
- Vehicle (Placebo Comparator): Participants in this group will be assigned a solution consisting of only the inactive ingredients in cromolyn sodium ophthalmic solution to apply to their entire face twice daily.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Cromolyn Sodium
  Other Names: Crolom
  Arms: Cromolyn
Drug: Normal Saline
  Other Names: 0.9% sodium chloride; NaCl
  Arms: Vehicle

SUMMARY:
This study is designed to investigate whether topical application of a cromolyn sodium solution is able to decrease the facial redness seen in patients with papulopustular rosacea. Previous work in the lab of Dr. Di Nardo on mice has suggested that cromolyn may be able to have this effect. The study will enroll a total of 10 patients. 5 will randomly be assigned to receive the cromolyn sodium solution, and the other 5 will be randomly assigned to receive the placebo solution. All participants will be instructed to apply their assigned solution twice daily to their face. Patients will return to the clinic 3, 6, and 8 weeks after the distribution of the solutions to measure the efficacy of their assigned solution.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or non-pregnant female, 18 - 80 years of age.
* Subjects willing and able to give informed consent.
* Subjects willing and able to comply with the requirements of the study.
* Subject has the clinical diagnosis of at least mild erythema.
* Subject has been on a stable dose for greater than 3 months of medications for treatment of concurrent medical condition (including oral contraceptive pills, vasodilators, adrenergic blocking agents) OR the investigator has determined that the medications are unlikely to affect the patient's rosacea and/or treatment during the study
* Subject is in general good health in the opinion of the investigator.

Exclusion Criteria:

* Subject has a diagnosis of Steroid Rosacea or Pyoderma Faciale (rosacea fulminans)
* Subject has a history of Carcinoid, Pheochromocytoma, Serotonin Syndrome or other systemic flushing causes.

Subject has used facial topical therapies (OTC drug products or prescription products) for any reason within the prior 28 days

* Subject has used systemic corticosteroid or systemic antibiotics (especially doxycycline, minocycline, tetracycline, metronidazole) within the prior 28 days.
* Subject has had laser or light-based treatment for rosacea within the prior 3 months.
* Subject has had systemic retinoids and retinoid derivatives over the past 6 months
* Subject has any history of renal or hepatic insufficiency.
* Subject has a known hypersensitivity or allergy to Cromolyn sodium or components of the vehicle.
* Subject is pregnant or lactating or planning a pregnancy during the duration of the study
* Subject has been treated with another investigational device or drug within 28 days prior to study enrollment or intends to participate in a clinical trial concurrent with this study
* Subject has clinically significant findings, medical history or conditions (other than rosacea), which in the opinion of the Investigator may compromise the study, treatment protocol, or safety of the patient or treatment allocation.

Subject has a known hypersensitivity or allergy to tape or other adhesive materials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Division of Dermatology, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cromolyn: Subjects in this arm will be asked to apply their assigned medication twice daily to their entire face. The medication they will be receiving is cromolyn sodium ophthalmic solution, 4%.
  Cromolyn Sodium
- Vehicle: Participants in this group will be assigned a solution consisting of only the inactive ingredients in cromolyn sodium ophthalmic solution to apply to their entire face twice daily.
  Normal Saline
Period: Overall Study
Arm/Group | Cromolyn | Vehicle
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cromolyn | Vehicle | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (5.2) | 62.6 (9.9) | 62.4 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Facial Erythema
Description: Facial erythema will be measured using the Clinician's Erythema Assessment(CEA) applied to 5 areas of the subject's face (chin, nose, glabella, left cheek, right cheek), as well as using measurements from a colorimeter applied to each of the 5 locations previous mentioned. Each area is rated from 0-4, where 4 represents the most facial erythema (worst outcome). The scores for the 5 locations are summed with a CEA total score scale of 0-20.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cromolyn | Vehicle
Number analyzed (Participants) | 5 | 5
score on a scale | 6.6 (1.9) | 6 (1.4)

2. Primary Outcome: Change in Facial Erythema
Description: We will measure participants' change in facial erythema over the course of the study. The change in facial erythema is measured as a difference between the final (8 weeks after baseline) and baseline visit of the sum of the CEA scores determined from the 5 designated locations (nose, glabella, left cheek, right cheek, and chin). The scale range from -20 to 20. A negative score indicates improvement of facial erythema from baseline to 8 weeks after baseline. A positive score indicates worsening of facial erythema from baseline to 8 weeks after baseline.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cromolyn | Vehicle
Number analyzed (Participants) | 5 | 5
score on a scale | -1.6 (2.6) | -0.8 (2.8)

3. Secondary Outcome: Matrix Metalloproteinase Activity Levels
Description: Tape stripping methods were used to isolate matrix metalloproteinase(MMP). Total-MMP activity was determined with total-MMP fluorogenic substrate (5 μM; Enzo Life Sciences), in protein extracts, and subsequently measuring activity (Vmax/sec) at a fluorescence excitation wavelength 328 nm and an emission wavelength of 400 nm in a fluorescence plate reader (Gemini EM microplate spectrofluorometer).
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: Vmax/sec
Arm/Group | Cromolyn | Vehicle
Number analyzed (Participants) | 5 | 5
Vmax/sec | 0.02 [0.0135 to 0.03] | 0.02 [0.013 to 0.025]

4. Secondary Outcome: Change in Matrix Metalloproteinase Activity
Description: We will compare subjects' matrix metalloproteinase activity levels at the beginning of the study (baseline) to those at the end of the study (8 weeks after baseline). Tape stripping methods were used to isolate matrix metalloproteinase(MMP). Total-MMP activity was determined with total-MMP fluorogenic substrate (5 μM; Enzo Life Sciences), in protein extracts, and subsequently measuring activity (Vmax/sec) at a fluorescence excitation wavelength 328 nm and an emission wavelength of 400 nm in a fluorescence plate reader (Gemini EM microplate spectrofluorometer).
Time Frame: Baseline and 8 weeks
Measure: Median (Inter-Quartile Range); unit: Vmax/sec
Arm/Group | Cromolyn | Vehicle
Number analyzed (Participants) | 5 | 5
Vmax/sec | -0.005 [-0.006 to 0] | 0.005 [0.004 to 0.008]

5. Other Pre Specified Outcome: Adverse Events
Description: Adverse events will be recorded at each visit and their likelihood to the study interventions will be recorded
Time Frame: Baseline, and then 3, 6 and 8 weeks after beginning study intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Cromolyn | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No